CLINICAL TRIAL: NCT01223924
Title: Randomized ，Placebo-controlled,Single-dose Escalation Trial of M2ES in Healthy Volunteer
Brief Title: Single-dose Escalation Trial of M2ES in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protgen Ltd (Industry)
Responsible Party: Guodong Chang, Protgen Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG-2008-1
Record Dates: First submitted 2010-10-09; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M2ES 7.5-90mg (Experimental): M2ES dose escalating
  Interventions: Drug: M2ES
- Placebo (Placebo Comparator): placebo contract
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — placebo
  Other Names: placebo conparator
  Arms: Placebo
Drug: M2ES — M2ES IV 7.5mg-90mg
  Other Names: M2ES esculating
  Arms: M2ES 7.5-90mg

SUMMARY:
This is a randomized double-blinded placebo-controlled，single-dose escalation trial in healthy volunteer.

DETAILED DESCRIPTION:
Randomized double-blinded placebo-controlled，single-dose escalation trial in health volunteer,to determine the safety and the max tolerate dose in health volunteer.

ELIGIBILITY:
Inclusion Criteria:

1. Physical and mental healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening.
2. 19 to 45 years of age.
3. Body mass index (19-25 kg/m2) ,the body weight ≥55kg for male subject,≥45kg for female.
4. Negative pregnant test, no menstrual period for female.
5. willing to comply with the protocol.

Exclusion Criteria:

1. Be allergic to endostatin
2. Have taken any drug during the last 2 weeks
3. Have Participated any clinical trail during the last 2 week
4. Cardiovasculre, respiratory, Liver, renal, gastro-intestinal hematologic endocrine and mental disease
5. HIV-1 infected
6. HBV, HBV infected ,Hepatitis B surface antigen positive

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine safety, toxicity and maxinum tolerable Dosage of M2ES injection in Safety and tolerability | 3 weeks
  To determine safety, toxicity and maxinum tolerable Dosage of M2ES injection in Subjects With Advanced Solid Tumors

SECONDARY OUTCOMES:
Pharmacokinetic (PK) behavior | 3 weeks
  Pharmacokinetic (PK) behavior of two different doses in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Ji JIANG, MD, Principal Investigator — Perking Union Medical College Hospital